CLINICAL TRIAL: NCT07223879
Title: Single Blind, Parallel Group Trial of Novel, On-Demand Virtual Reality to Amplify Practice Efficacy (NO VAPE) Added to Cognitive Behavioral Therapy for Nicotine Vaping Cessation
Brief Title: Trial of Novel, On-Demand Virtual Reality to Amplify Practice Efficacy (NO VAPE) Added to Cognitive Behavioral Therapy for Nicotine Vaping Cessation
Acronym: NO VAPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles River Analytics (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00087216; 4R44DA059018-02 (NIH)
Record Dates: First submitted 2025-10-24; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: NO VAPE + 12 Weeks of Standard CBT; Sham NO VAPE + 12 Weeks Standard CBT

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NO VAPE + 12 weeks CBT (Active Comparator): The experimental group will receive the following over a 12-week period: NO VAPE (VR app) combined with the MGH 12-session remote behavioral vaping cessation support program for vaping cessation.
  Interventions: Behavioral: NO VAPE VR app with CBT-embedded content with a 12-session individual CBT treatment program
- Sham NO VAPE + 12 weeks CBT (Sham Comparator): The control group will receive a sham NO VAPE (VR app) combined with the MGH 12-session remote behavioral vaping cessation support program.
  Interventions: Behavioral: Sham VR app without CBT-embedded content with a 12-session individual CBT treatment program

INTERVENTIONS:
Behavioral: NO VAPE VR app with CBT-embedded content with a 12-session individual CBT treatment program — The control group will receive a sham NO VAPE (VR app) combined with the MGH 12-session remote behavioral vaping cessation support program.
  Arms: NO VAPE + 12 weeks CBT
Behavioral: Sham VR app without CBT-embedded content with a 12-session individual CBT treatment program — The control group will receive a sham NO VAPE (VR app) combined with the MGH 12-session remote behavioral vaping cessation support program.
  Arms: Sham NO VAPE + 12 weeks CBT

SUMMARY:
3. General Description of Study Design

The proposed study will evaluate the effect of adding a VR app with CBT-embedded content to a 12-session individual CBT treatment program. Investigators propose a prospective, randomized, single-blind, trial with 90 individuals aged 16 years and over who vape nicotine at least weekly for three months, and wish to quit vaping within the next month. Subjects will be randomly assigned to either the experimental (NO VAPE + CBT) or control group (sham NO VAPE + CBT) for 12 weeks. The study will use a double blind design where both subjects and investigators and outcome assessors will be masked to subjects' group assignments. The experimental group will receive the following over a 12-week period: NO VAPE (VR app) combined with the MGH 12-session remote behavioral vaping cessation support program for vaping cessation. The control group will receive a sham NO VAPE (VR app) combined with the MGH 12-session remote behavioral vaping cessation support program. The VR app will be used at home by participants in between CBT session visits. Participants will also briefly report their CBT skills practice using the MyCap smartphone app. Participants will be assigned randomly to the experimental or control group in a 1:1 ratio, with randomization blocks of 6, stratified by no/mild nicotine dependence (Electronic Cigarette Dependence Index [ECDI] score 0-8) or moderate/high nicotine dependence (ECDI score 9 or higher) in a prospective trial in people age 16 and over, who use vaped nicotine regularly and wish to quit vaping.

The primary outcome is self-reported time spent in CBT skills practice per week. Groups will be compared on mean number of days and duration of self-reported CBT skill practice per week over the 12-week treatment period.

Secondary outcomes are: tolerability and feasibility of the NO VAPE virtual reality (VR) vaping cessation tool, which will be assessed by the following self-reported ratings in both groups: a) average CBT session attendance weekly, b) satisfaction ratings, c) adverse events; and by the following self-reported ratings d) self-ratings of the virtual reality application usability, e) engagement, f) presence, and g) simulator cyber sickness.

Exploratory outcomes are: 1) biochemically verified 7-day point prevalence vaping abstinence at week 12, and 2) 4-week biochemically verified continuous abstinence from weeks 9-12.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Report of nicotine vaping at least weekly for the prior ≥ 3 months
* Self-report of not smoking tobacco regularly at enrollment (tobacco smoking on <8 of the past 30 days)
* Report motivation to quit vaping in the next 30 days
* Own or are willing to use a Meta Quest VR headset
* Vision corrected to within 20/50 bilaterally
* Access to a mobile device to complete daily survey assessments
* If age is greater than or equal to 18 years: Competent and willing to provide written informed consent
* If age is less than 18 years: Competent and willing to provide written informed assent AND have a parent/legal guardian who is competent and willing to provide written informed consent

Exclusion Criteria:

* Individuals at greater risk of harm from virtual reality side effects, such as a history of motion sickness, history of migraines or severe headaches, history of vertigo, epilepsy or neurological conditions where visual stimuli may trigger seizures or other issues (excludes history of febrile seizures), or self-report of pregnancy, recent concussion, or other conditions that increase risks of dizziness, nausea, or headaches
* Evidence of active problem substance use severe enough, in the investigator's opinion, to compromise ability to safely participate
* Unwilling to provide saliva or urine samples
* Any condition or situation that would, in the investigator's opinion, make it unlikely that the participant could adhere safely to the study protocol
* Individuals who are under the legal protection of the government or state (Wards of the State)
* Inability to understand study procedures, read, and write in English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Difference in CBT sessions attended | 12 Weeks
  We will evaluate the number of CBT sessions attended across the 12 weeks
Time spent practicing CBT skills | Weeks 1-12
  We time spent practicing CBT between sessions in minutes. The app collects data automatically on how much time is spent using it, and how much time is spent within each environment.

SECONDARY OUTCOMES:
Change in craving | Weeks 1-12
  We will measure changes in craving at enrollment and weekly using a brief, 10-item, valid and reliable measure of vaping craving that queries desire and intent to vape and anticipation of positive outcomes related to e-cigarette use.
Change in withdrawal symptoms | Weeks 1-12
  We will measure changes in withdrawal symptoms using the Minnesota Nicotine Withdrawal Scale (MNWS)
Change in severity of tobacco use disorder (TUD) | Week 12
  We will evaluate the impact of the intervention on reducing the severity of tobacco use disorder (TUD). Severity of TUD is operationalized as Electronic Cigarette Dependence Index (ECDI; Foulds et al., 2015) total score, (range 0-20).

OTHER OUTCOMES:
7-Day Point Prevalence Vaping Abstinence | week 12
  Exploratory outcome 1 is biochemically verified 7-day point prevalence vaping abstinence at week 12.
4-Week Vaping Abstinence | weeks 9-12
  Exploratory outcome 2 is 4-week biochemically verified continuous abstinence from weeks 9-12.

IPD SHARING:
Plan to Share IPD: Yes
All Deidentified IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Feb 2029
Access Criteria: They must request access through Charles River Analytics.

REFERENCES:
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Kennedy RS, Lane NE, Berbaum KS, Lilienthal MG. Simulator Sickness Questionnaire: An Enhanced Method for Quantifying Simulator Sickness. The International Journal of Aviation Psychology. 1993/07/01 1993;3(3):203-220. doi:10.1207/s15327108ijap0303_3
- [Background] Witmer BG, Singer MJ. Measuring Presence in Virtual Environments: A Presence Questionnaire. Presence: Teleoperators and Virtual Environments. 1998;7(3):225-240. doi:10.1162/105474698565686
- [Background] Lin JJW, Duh HBL, Parker DE, Abi-Rached H, Furness TA. Effects of field of view on presence, enjoyment, memory, and simulator sickness in a virtual environment. 2002:164-171.
- [Background] Schuster RM, Cather C, Pachas GN, Nielsen L, Iroegbulem V, Dufour J, Potter K, Levy S, Gray KM, Evins AE. A randomized controlled trial of varenicline and brief behavioral counseling delivered by lay counselors for adolescent vaping cessation: Study protocol. Front Psychiatry. 2023 Mar 15;14:1083791. doi: 10.3389/fpsyt.2023.1083791. eCollection 2023. PMID 37009114
- [Background] Meta. This is Meta Quest. Accessed 03/05/2025, 2025. https://www.meta.com/quest/?srsltid=AfmBOoojbfuf4Ht9amTr-QDOGrgC5wz7RHJ80CTGLUZ4bQ0IKlyr_V8w
- [Background] Hughes JR, Hatsukami D. Signs and symptoms of tobacco withdrawal. Arch Gen Psychiatry. 1986 Mar;43(3):289-94. doi: 10.1001/archpsyc.1986.01800030107013. PMID 3954551
- [Background] Dowd AN, Motschman CA, Tiffany ST. Development and Validation of the Questionnaire of Vaping Craving. Nicotine Tob Res. 2019 Jan 1;21(1):63-70. doi: 10.1093/ntr/nty046. PMID 29546379
- [Background] Piper ME, Baker TB, Benowitz NL, Smith SS, Jorenby DE. E-cigarette Dependence Measures in Dual Users: Reliability and Relations With Dependence Criteria and E-cigarette Cessation. Nicotine Tob Res. 2020 Apr 21;22(5):756-763. doi: 10.1093/ntr/ntz040. PMID 30874804
- [Background] Adamson SJ, Kay-Lambkin FJ, Baker AL, Lewin TJ, Thornton L, Kelly BJ, Sellman JD. An improved brief measure of cannabis misuse: the Cannabis Use Disorders Identification Test-Revised (CUDIT-R). Drug Alcohol Depend. 2010 Jul 1;110(1-2):137-43. doi: 10.1016/j.drugalcdep.2010.02.017. Epub 2010 Mar 26. PMID 20347232
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Robinson SM, Sobell LC, Sobell MB, Leo GI. Reliability of the Timeline Followback for cocaine, cannabis, and cigarette use. Psychol Addict Behav. 2014 Mar;28(1):154-62. doi: 10.1037/a0030992. Epub 2012 Dec 31. PMID 23276315
- [Background] Wienrich C, Döllinger N, Hein R. Behavioral Framework of Immersive Technologies (BehaveFIT): How and Why Virtual Reality can Support Behavioral Change Processes. Hypothesis and Theory. Frontiers in Virtual Reality. 2021-June-24 2021;2doi:10.3389/frvir.2021.627194
- [Background] Okpako T, Kale D, Perski O, Brown J. Prevalence and characteristics of smokers interested in using virtual reality for encouraging smoking cessation: a representative population survey in Great Britain. BMC Digital Health. 2024/11/12 2024;2(1):79. doi:10.1186/s44247-024-00136-2
- [Background] Pericot-Valverde I, Secades-Villa R, Gutierrez-Maldonado J, Garcia-Rodriguez O. Effects of systematic cue exposure through virtual reality on cigarette craving. Nicotine Tob Res. 2014 Nov;16(11):1470-7. doi: 10.1093/ntr/ntu104. Epub 2014 Jun 23. PMID 24962558
- [Background] Pericot-Valverde I, Secades-Villa R, Gutierrez-Maldonado J. A randomized clinical trial of cue exposure treatment through virtual reality for smoking cessation. J Subst Abuse Treat. 2019 Jan;96:26-32. doi: 10.1016/j.jsat.2018.10.003. Epub 2018 Oct 16. PMID 30466545
- [Background] Pericot-Valverde I, Garcia-Rodriguez O, Gutierrez-Maldonado J, Ferrer-Garcia M, Secades-Villa R. Evolution of smoking urge during exposure through virtual reality. Stud Health Technol Inform. 2011;167:74-9. PMID 21685645
- [Background] Mayer M, Reyes-Guzman C, Grana R, Choi K, Freedman ND. Demographic Characteristics, Cigarette Smoking, and e-Cigarette Use Among US Adults. JAMA Netw Open. 2020 Oct 1;3(10):e2020694. doi: 10.1001/jamanetworkopen.2020.20694. PMID 33048127
- [Background] Wang P, Ai X, Zhang X, Ma F, Zhuang Y, Wang S. Evaluating virtual reality technology in psychotherapy: impacts on anxiety, depression, and ADHD. Front Psychiatry. 2024 Dec 18;15:1480788. doi: 10.3389/fpsyt.2024.1480788. eCollection 2024. PMID 39744548
- [Background] Lindner P. Better, Virtually: the Past, Present, and Future of Virtual Reality Cognitive Behavior Therapy. International Journal of Cognitive Therapy. 2021/03/01 2021;14(1):23-46. doi:10.1007/s41811-020-00090-7
- [Background] Keijsers M, Vega-Corredor MC, Tomintz M, Hoermann S. Virtual Reality Technology Use in Cigarette Craving and Smoking Interventions (I "Virtually" Quit): Systematic Review. J Med Internet Res. 2021 Sep 17;23(9):e24307. doi: 10.2196/24307. PMID 34533471
- [Background] Milkowski M, Olesk J, Asfura DM, et al. Youth Vaping in the Digital Age: A Systematic Review of Technological Interventions for Prevention and Cessation. presented at: Companion Proceedings of the 2025 ACM International Conference on Supporting Group Work; 2025; Hilton Head, New Jersey, USA. https://doi.org/10.1145/3688828.3699642
- [Background] Obisesan OH, Osei AD, Uddin SMI, Dzaye O, Mirbolouk M, Stokes A, Blaha MJ. Trends in e-Cigarette Use in Adults in the United States, 2016-2018. JAMA Intern Med. 2020 Oct 1;180(10):1394-1398. doi: 10.1001/jamainternmed.2020.2817. PMID 32897288
- [Background] Vahratian A, Briones EM, Jamal A, Marynak KL. Electronic Cigarette Use Among Adults in the United States, 2019-2023. NCHS Data Brief. 2025 Jan;(524):CS356607. doi: 10.15620/cdc/174583. PMID 40036117
- [Background] Bandi P, Star J, Minihan AK, Patel M, Nargis N, Jemal A. Changes in E-Cigarette Use Among U.S. Adults, 2019-2021. Am J Prev Med. 2023 Aug;65(2):322-326. doi: 10.1016/j.amepre.2023.02.026. Epub 2023 Apr 18. PMID 37479423